CLINICAL TRIAL: NCT03675308
Title: A Phase 3, Randomized, Double-Blind, Study Comparing Risankizumab to Placebo in Subjects With Active Psoriatic Arthritis (PsA) Who Have a History of Inadequate Response to or Intolerance to at Least One Disease Modifying Anti-Rheumatic Drug (DMARD) Therapy (KEEPsAKE 1)
Brief Title: A Study Comparing Risankizumab to Placebo in Participants With Active Psoriatic Arthritis (PsA) Who Have a History of Inadequate Response to or Intolerance to at Least One Disease Modifying Anti-Rheumatic Drug (DMARD) Therapy
Acronym: KEEPsAKE 1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M16-011; 2017-002465-22 (EudraCT Number)
Record Dates: First submitted 2018-09-12; First posted 2018-09-18 (Actual); Results first posted 2022-02-24 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants randomized to receive double-blind placebo at Week 0, Week 4, and Week 16 in Period 1. At Week 24 participants will receive 150 mg risankizumab followed by open-label 150 mg risankizumab at Week 28, and every 12 weeks thereafter in Period 2 until the final dosing time point at Week 316.
  Interventions: Biological: Placebo; Biological: Risankizumab
- Risankizumab (Experimental): Participants randomized to receive 150 mg risankizumab administered by subcutaneous injection at Week 0, Week 4, and Week 16 in Period 1. At Week 24 participants will receive blinded placebo followed by open-label 150 mg risankizumab at Week 28, and every 12 weeks thereafter in Period 2 until the final dosing time point at Week 316.
  Interventions: Biological: Placebo; Biological: Risankizumab

INTERVENTIONS:
Biological: Placebo — Placebo for risankizumab administered by subcutaneous injection
Biological: Risankizumab — Risankizumab administered by subcutaneous injection
  Other Names: ABBV-066; BI 655066; SKYRIZI

SUMMARY:
The purpose of this study is to compare the safety and efficacy of risankizumab versus placebo in participants with moderately to severely active psoriatic arthritis (PsA).

DETAILED DESCRIPTION:
The study consists of a Screening Period (approximately 35 days), Period 1, Period 2, and a 20-week Follow-up Period. Period 1 is a 24-week randomized, double-blind, placebo-controlled, parallel-group treatment period. Period 2 is the long-term treatment period and starts at Week 24. To maintain the blind to the original treatment allocation, treatment at the Week 24 Visit is blinded: participants randomized to placebo receive blinded risankizumab 150 mg, and participants randomized to risankizumab receive blinded placebo. At Week 28 and for the remaining dosing visits (to Week 316), all participants are to receive open-label risankizumab 150 mg every 12 weeks. Participants will remain blinded to the original randomization allocation for the duration of the study. The total study duration is 336 weeks including a telephone call 140 days (20 weeks) after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PsA with symptom onset at least 6 months prior to the Screening Visit and fulfillment of the Classification Criteria for PsA (CASPAR) at the Screening Visit.
* Participant has active disease at Baseline defined as ≥ 5 tender joints (based on 68 joint counts) and ≥ 5 swollen joints (based on 66 joint counts)
* Diagnosis of active plaque psoriasis with at least one psoriatic plaque of ≥ 2 cm diameter or nail changes consistent with psoriasis at Screening Visit.
* Participant has demonstrated an inadequate response or intolerance to or contraindication for conventional synthetic disease modifying anti-rheumatic drugs (csDMARD) therapy(ies).
* Presence of either at Screening:

  * ≥ 1 erosion on radiograph as determined by central imaging review or;
  * High sensitivity C-reactive protein (hsCRP) ≥ 3.0 mg/L.

Exclusion Criteria:

* Participant is considered by investigator, for any reason, to be an unsuitable candidate for the study.
* Participant has a known hypersensitivity to risankizumab.
* Participant has previous treatment with biologic agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 964 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2026-09-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (256):
- United States (59):
  - Pinnacle Research Group /ID# 167955, Anniston, Alabama
  - Sun Valley Arthritis Center Ltd. /ID# 200270, Peoria, Arizona
  - AZ Arthritis and Rheumotology Research, PLLC /ID# 209873, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC /ID# 209875, Tucson, Arizona
  - Southern Arizona VA Health Care System /ID# 209247, Tucson, Arizona
  - Arthritis and Rheumatism Associates /ID# 209882, Jonesboro, Arkansas
  - Valerius Medical Group & Research Center /ID# 207428, Los Alamitos, California
  - Rheumatology Center of San Diego /ID# 201642, San Diego, California
  - Inland Rheum Clin Trials Inc. /ID# 201641, Upland, California
  - Medvin Clinical Research /ID# 211127, Whittier, California
  - New England Research Associates, LLC /ID# 207237, Bridgeport, Connecticut
  - Danbury Clinical Research, LLC /ID# 209517, Danbury, Connecticut
  - Arthritis & Osteoporosis Center /ID# 207236, Hamden, Connecticut
  - Arthritis & Rheumatic Disease Specialties /ID# 210802, Aventura, Florida
  - Rheumatology Associates of South Florida (RASF) - Clinical Research /ID# 211099, Boca Raton, Florida
  - SIMED Health, LLC /ID# 207461, Gainesville, Florida
  - Sweet Hope Research Specialty Inc /ID# 209393, Hialeah, Florida
  - Jacksonville Center for Clinical Research /ID# 209876, Jacksonville, Florida
  - Rheum Assoc of Central FL /ID# 201622, Orlando, Florida
  - HMD Research LLC /ID# 208427, Orlando, Florida
  - IRIS Research and Development, LLC /ID# 208955, Plantation, Florida
  - ForCare Clinical Research /ID# 168034, Tampa, Florida
  - Arthritis and Rheumatology /ID# 168046, Atlanta, Georgia
  - Affinity Clinical Research /ID# 210816, Oak Brook, Illinois
  - OrthoIllinois /ID# 205300, Rockford, Illinois
  - Springfield Clinic /ID# 200244, Springfield, Illinois
  - Klein and Associates MD /ID# 169483, Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research /ID# 168017, Wheaton, Maryland
  - Clinical Pharmacology Study Gr /ID# 168019, Worcester, Massachusetts
  - Advanced Rheumatology, PC /ID# 168042, Lansing, Michigan
  - June DO, PC /ID# 208915, Lansing, Michigan
  - St. Paul Rheumatology /ID# 208471, Eagan, Minnesota
  - Logan Health Research /ID# 213707, Kalispell, Montana
  - Physician Research Collaboration, LLC /ID# 208670, Lincoln, Nebraska
  - Center for Rheumatology LLP /ID# 207313, Albany, New York
  - NYU Langone Ambulatory Care Brooklyn Heights /ID# 207310, Brooklyn, New York
  - Joint & Muscle Research Instit /ID# 208620, Charlotte, North Carolina
  - Medication Management, LLC /ID# 211734, Greensboro, North Carolina
  - Coastal Carolina Health Care /ID# 208619, New Bern, North Carolina
  - Velocity Clinical Research /ID# 200452, Blue Ash, Ohio
  - Marietta Memorial Hospital /ID# 210179, Marietta, Ohio
  - Paramount Medical Research Con /ID# 201583, Middleburg Heights, Ohio
  - STAT Research, Inc. /ID# 213805, Springboro, Ohio
  - Health Research of Oklahoma /ID# 168027, Oklahoma City, Oklahoma
  - Altoona Ctr Clinical Res /ID# 168037, Duncansville, Pennsylvania
  - Allegheny Health Network Research Institute /ID# 210349, Pittsburgh, Pennsylvania
  - Clinical Research Ctr Reading /ID# 168070, Wyomissing, Pennsylvania
  - Nashville Arthritis and Rheumatology /ID# 168069, Nashville, Tennessee
  - Amarillo Ctr for Clin Research /ID# 208347, Amarillo, Texas
  - Precision Comprehensive Clinical Research Solutions /ID# 208386, Colleyville, Texas
  - Dallas VA Medical Center /ID# 208389, Dallas, Texas
  - Precision Comprehensive Clinical Research Solutions /ID# 210597, Fort Worth, Texas
  - Advanced Rheumatology of Houston /ID# 208354, The Woodlands, Texas
  - DM Clinical Research /ID# 208351, Tomball, Texas
  - Kadlec Clinic Rheumatology /ID# 207969, Kennewick, Washington
  - Rheumatology and Pulmonary Clinic /ID# 200446, Beckley, West Virginia
  - Aurora Rheumatology and Immunotherapy Center /ID# 168066, Franklin, Wisconsin
  - Holy Family Memorial, Inc. /ID# 209387, Manitowoc, Wisconsin
  - Gundersen Clinic, Ltd /ID# 209459, Onalaska, Wisconsin
- Argentina (12):
  - Framingham Centro Medico /ID# 210409, La Plata, Buenos Aires
  - Hospital General de Agudos J. M. Ramos Mejia /ID# 169164, Buenos Aires, Ciuadad Autonoma de Buenos Aires
  - Hospital Italiano de Buenos Aires /ID# 208474, Ciudad Autonoma Buenos Aires, Ciuadad Autonoma de Buenos Aires
  - DOM Centro de Reumatologia /ID# 208479, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Fundacion CIDEA /ID# 210494, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich /ID# 211622, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Centro de Enfermedades del Hígado y Aparato Digestivo /ID# 169163, Rosario, Santa Fe Province
  - Instituto CAICI /ID# 169168, Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia /ID# 208343, San Miguel de Tucumán, Tucumán Province
  - Duplicate_Inst de Rehab Psicofisica /ID# 214681, Buenos Aires
  - Duplicate_Hospital Privado Univesitario /ID# 211623, Córdoba
  - Cimer /Id# 169167, San Miguel de Tucumán
- Australia (7):
  - The Canberra Hospital /ID# 207592, Garran, Australian Capital Territory
  - Royal Brisbane and Women's Hospital /ID# 212785, Herston, Queensland
  - Rheumatology Research Unit Sunshine Coast /ID# 207200, Maroochydore, Queensland
  - Griffith University /ID# 207505, Southport, Queensland
  - Flinders Medical Centre /ID# 210562, Bedford Park, South Australia
  - Emeritus Research /ID# 207202, Camberwell, Victoria
  - Monash Medical Centre /ID# 208034, Clayton, Victoria
- Belgium (3):
  - Duplicate_UZ Ghent /ID# 210036, Ghent, Oost-Vlaanderen
  - ReumaClinic /ID# 208213, Genk
  - ZNA - Jan Palfijn /ID# 208212, Merksem
- Bosnia and Herzegovina (4):
  - University Clinical Centre of the Republic of Srpska /ID# 208268, Banja Luka, Republika Srpska
  - University Clinical Centre of the Republic of Srpska /ID# 208269, Banja Luka, Republika Srpska
  - University Clinical Centre of the Republic of Srpska /ID# 210047, Banja Luka, Republika Srpska
  - Clinical Center University of Sarajevo /ID# 208272, Sarajevo
- Brazil (5):
  - SER - Serviços Especializados em Reumatologia /ID# 207489, Salvador, Estado de Bahia
  - CMiP - Centro Mineiro de Pesquisa Ltda - ME /ID# 207496, Juiz de Fora, Minas Gerais
  - EDUMED Educacao em Saude S/S L /ID# 207488, Curitiba, Paraná
  - LMK Sevicos Medicos S/S /ID# 207491, Porto Alegre, Rio Grande do Sul
  - CPCLIN - Centro de Pesquisas Clínicas /ID# 207493, São Paulo
- Bulgaria (4):
  - Medical center Medconsult /ID# 211399, Pleven
  - Medical center Excelsior /ID# 167741, Sofia
  - Diagnostic consultative center 17 Sofia /ID# 210506, Sofia
  - Military Medical Academy Multiprofile Hospital /ID# 210829, Sofia
- Canada (7):
  - Percuro Clinical Research, Ltd /ID# 169601, Victoria, British Columbia
  - Manitoba Clinic /ID# 206819, Winnipeg, Manitoba
  - CIADS Research Co Ltd /ID# 169600, Winnipeg, Manitoba
  - SKIN Centre for Dermatology /ID# 169604, Peterborough, Ontario
  - K. Papp Clinical Research /ID# 169603, Waterloo, Ontario
  - Groupe de Recherche en Maladies Osseuses Inc /ID# 169598, Sainte-Foy, Quebec
  - Dr. Latha Naik /ID# 212188, Saskatoon, Saskatchewan
- Chile (3):
  - CTR Estudios Clinicos /ID# 208166, Providencia
  - Centro Internacional de Estudios Clinicos /ID# 209908, Santiago
  - Clinica Dermacross S.A /ID# 208163, Vitacura Santiago
- Croatia (7):
  - Poliklinika Repromed /ID# 208628, Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 210965, Zagreb, City of Zagreb
  - UHC Osijek /ID# 208623, Osijek, County of Osijek-Baranja
  - Klinicki bolnicki centar Rijeka /ID# 208621, Rijeka, Primorje-Gorski Kotar County
  - Klinicki bolnicki centar Split /ID# 208626, Split, Split-Dalmatia County
  - Medical Center Kuna-Peric /ID# 208047, Zagreb
  - Poliklinika Bonifarm /ID# 208750, Zagreb
- Czechia (5):
  - Revmacentrum MUDr. Mostera, s.r.o. /ID# 209025, Brno
  - PV MEDICAL Services s.r.o. /ID# 210222, Prague
  - MUDr. Zuzana Stejfova - revmatologicka ambulance /ID# 209027, Prague
  - Affidea Praha s.r.o. /ID# 210223, Prague
  - MEDICAL PLUS, s.r.o. /ID# 210439, Uherské Hradiště
- Denmark (2):
  - Bispebjerg and Frederiksberg Hospital /ID# 207576, Frederiksberg, Capital Region
  - Aarhus University Hospital /ID# 168761, Aarhus C, Central Jutland
- Estonia (3):
  - North Estonia Medical Centre /ID# 208325, Mustamäe, Harju
  - Innomedica /ID# 211416, Tallinn, Harju
  - MediTrials /ID# 207816, Tartu, Tartu
- Finland (3):
  - Helsinki University Hospital /ID# 207724, Helsinki, Uusimaa
  - Ite Pihlajanlinna Kuopio /ID# 208322, Kuopio
  - Turku University Hospital /ID# 207726, Turku
- Germany (4):
  - Rheumazentrum Ruhrgebiet /ID# 207216, Herne, North Rhine-Westphalia
  - Immanuel Krankenhaus Berlin /ID# 207218, Buch
  - Center of Innovative Diagnostics and Therapeutics (CIRI GmbH) /ID# 209483, Frankfurt
  - MVZ Rheumatologie und Autoimmunmedizin Hamburg GmbH /ID# 209484, Hamburg
- Greece (5):
  - General Hospital Asklepieio Voulas /ID# 212956, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 206839, Heraklion, Crete
  - 424 General MILITARY Hospital /ID# 210974, Efkarpia (Thessalonikis), Thessaloniki
  - Naval Hospital of Athens /ID# 206838, Athens
  - Olympion General Clinic SA /ID# 207048, Pátrai
- Israel (5):
  - Sheba Medical Center /ID# 207474, Ramat Gan, Tel Aviv
  - Barzilai Medical Center /ID# 207476, Ashkelon
  - Rambam Health Care Campus /ID# 208170, Haifa
  - Meir Medical Center /ID# 207473, Kfar Saba
  - Rabin Medical Center /ID# 207475, Petah Tikva
- Italy (5):
  - Duplicate_Azienda Ospedaliero-Universitaria Policlinico di Modena /ID# 207799, Modena, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona /ID# 207269, Ancona
  - A.O.U. Policlinico G. Rodolico S.Marco - Presidio San Marco /ID# 207795, Catania
  - Duplicate_Policlinico Univ Tor Vergata /ID# 207271, Rome
  - Azienda Ospedaliera Universitaria di Verona/Ospedale Borgo Roma /ID# 207265, Verona
- Latvia (5):
  - M & M Centrs LTD /ID# 208733, Ādaži
  - D.Saulites-Kandevicas PP in Cardiology and Rheumatology /ID# 207224, Liepāja
  - Pauls Stradins Clinical University Hospital /ID# 207220, Riga
  - Clinic ORTO /ID# 216218, Riga
  - Riga East Clinical University Hospital /ID# 207223, Riga
- Lithuania (4):
  - VAKK Dr. Kilda's Clinic /ID# 207330, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 207331, Kaunas
  - Klaipeda University Hospital /ID# 207329, Klaipėda
  - Republican Siauliai hospital /ID# 207328, Šiauliai
- Malaysia (4):
  - Hospital Tuanku Jaafar /ID# 207919, Seremban, Negeri Sembilan
  - Hospital Raja Permaisuri Bainun /ID# 207920, Ipoh, Perak
  - Hospital Selayang /ID# 208938, Batu Caves, Selangor
  - University Malaya Med Ctr /ID# 208937, Kuala Lumpur
- Mexico (6):
  - Centro Integral en Reumatologia S.A de C.V /ID# 208346, Guadalajara, Jalisco
  - CINTRE, Centro de Investigación y Tratamiento Reumatológico SC /ID# 208331, Mexico City, Mexico City
  - Eukarya PharmaSite, SC /ID# 208431, Monterrey, Nuevo León
  - Centro Peninsular de Investigación Clínica SCP /ID# 208345, Colonia Centro, Yucatán
  - Hospital General Regional No. 1 Dr. Carlos Mac Gregor Sánchez Navarro /ID# 210835, Mexico City
  - RM Pharma Specialists S.A de C.V /ID# 208330, Mexico City
- Netherlands (3):
  - Antonius Ziekenhuis /ID# 208587, Sneek, Provincie Friesland
  - Universitair Medisch Centrum Groningen /ID# 208580, Groningen
  - Medisch Centrum Leeuwarden /ID# 168453, Leeuwarden
- New Zealand (3):
  - Middlemore Clinical Trials /ID# 213256, Papatoetoe, Auckland
  - Waikato Hospital /ID# 213257, Hamilton, Waikato Region
  - CGM Research Trust /ID# 210498, Burwood
- Poland (9):
  - Spolka Lekarzy INTERCOR /ID# 210191, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Nasz Lekarz Przychodnie Medyczne /ID# 216176, Torun, Kuyavian-Pomeranian Voivodeship
  - Malopolskie Centrum Kliniczne /ID# 208007, Krakow, Lesser Poland Voivodeship
  - McBk Sc /Id# 209132, Grodzisk Mazowiecki, Masovian Voivodeship
  - Centrum Medyczne Reuma Park w Warszawie /ID# 210352, Warsaw, Masovian Voivodeship
  - Osteo-Medic S.C. /ID# 208008, Bialystok, Podlaskie Voivodeship
  - ClinicMed Daniluk, Nowak Sp.j. /ID# 210824, Bialystok, Podlaskie Voivodeship
  - Centrum Kliniczno-Badawcze /ID# 208010, Elblag, Warmian-Masurian Voivodeship
  - ETYKA-Osrodek Badan Klinicznych /ID# 216241, Olsztyn, Warmian-Masurian Voivodeship
- Portugal (6):
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, EPE /ID# 208145, Vila Nova de Gaia, Porto District
  - Unidade Local de Saúde do Alto Minho, EPE - Hospital Conde de Bertiandos /ID# 208147, Ponte de Lima, Viana do Castelo District
  - Centro Hospitalar do Baixo Vouga /ID# 215979, Aveiro
  - CCA Braga - Hospital de Braga /ID# 208146, Braga
  - Instituto Português De Reumatologia /ID# 208149, Lisbon
  - Centro Hospitalar Universitário de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 208148, Lisbon
- Mindful Medical Research /ID# 211129, San Juan, Puerto Rico
- Romania (4):
  - Cabinet Medical Dr Triff Carina /Id# 207528, Timișoara, Timiș County
  - Spitalul Clinic Sf. Maria /ID# 210054, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj -Napoca /ID# 207340, Cluj-Napoca
  - Spitalul Clinic de Recuperare Iasi /ID# 207371, Iași
- Russia (8):
  - LLC Family Outpatient Clinic № /ID# 169510, Korolev, Moscow
  - Research Institute of Rheumatology named after V.A. Nasonova /ID# 207643, Moscow, Moscow
  - LLC Medical Center /ID# 169516, Novosibirsk, Novosibirsk Oblast
  - Nort-Western State Medical University n.a. Mechnikov /ID# 207641, Saint Petersburg, Sankt-Peterburg
  - Kazan State Medical University /ID# 169511, Kazan', Tatarstan, Respublika
  - Federal Center for Brain and Neurotechnology /ID# 207646, Moscow
  - Perm Regional Clinical Hospital /ID# 207642, Perm
  - Ulyanovsk Regional Clinical Hospital /ID# 169515, Ulyanovsk
- Serbia (7):
  - Institute for Rheumatology /ID# 168194, Belgrade, Beograd
  - Institute for Rheumatology /ID# 168197, Belgrade, Beograd
  - Institute for Rheumatology /ID# 168198, Belgrade, Beograd
  - Institute for Rheumatology /ID# 168199, Belgrade, Beograd
  - Military Medical Academy /ID# 168218, Belgrade, Beograd
  - Special Hospital for Rheuma /ID# 168255, Novi Sad, Vojvodina
  - Special Hospital for Rheuma /ID# 210284, Novi Sad, Vojvodina
- Singapore (3):
  - National University Hospital /ID# 208599, Singapore
  - Singapore General Hospital /ID# 207917, Singapore
  - Changi General Hospital /ID# 208965, Singapore
- Slovakia (5):
  - REUMA-GLOBAL, s.r.o. /ID# 208017, Biely Kostol
  - MEDMAN s.r.o. /ID# 208018, Martin
  - Reum.hapi s.r.o. /ID# 208016, Nové Mesto nad Váhom
  - Thermium s.r.o. /ID# 208015, Piešťany
  - REUMAMED POPRAD s.r.o. /ID# 208407, Poprad
- South Africa (6):
  - Dr Jenny Potts /ID# 168691, Port Elizabeth, Eastern Cape
  - University of Pretoria /ID# 167621, Pretoria, Gauteng
  - Dr Elsa van Duuren /ID# 207577, Pretoria, Gauteng
  - Arthritis Clinical Research Trials /ID# 167625, Cape Town, Western Cape
  - Synexus Helderberg Clinical Research Centre /ID# 210891, Somerset West, Western Cape
  - Winelands Medical Research Centre /ID# 167629, Stellenbosch, Western Cape
- South Korea (3):
  - Hanyang University Seoul Hospital /ID# 209263, Seoul, Seoul Teugbyeolsi
  - Duplicate_Konkuk University Medical Ctr /ID# 207509, Seoul, Seoul Teugbyeolsi
  - Kyungpook National Univ Hosp /ID# 207408, Daegu
- Spain (8):
  - Hospital Universitario Germans Trias i Pujol /ID# 208543, Badalona, Barcelona
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 207830, Sabadell, Barcelona
  - Hospital Universitario A Coruna - CHUAC /ID# 207826, A Coruña
  - Hospital Universitario Torrecardenas /ID# 212716, Almería
  - Hospital Parc de Salut del Mar /ID# 209698, Barcelona
  - Hospital Clinico Universitario San Carlos /ID# 207832, Madrid
  - Hospital Universitario 12 de Octubre /ID# 207827, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 207831, Valencia
- Sweden (6):
  - Skane University hospital /ID# 210070, Malmo, Skåne County
  - Falu Lasarett /ID# 210322, Falun
  - Duplicate_Karolinska Univ Sjukhuset /ID# 208175, Solna
  - Uppsala University Hospital /ID# 207944, Uppsala
  - Duplicate_Vastmanlands Sjukhus /ID# 207943, Västerås
  - Orebro Universitetssjukhuset /ID# 207948, Örebro, Örebro County
- Taiwan (3):
  - Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation /ID# 207567, Chiayi City
  - Chung Shan Medical University Hospital /ID# 207257, Taichung
  - Linkou Chang Gung Memorial Ho /ID# 207255, Taoyuan
- Ukraine (12):
  - State Institution L. T. Malaya Therapy National Institution of NAMS of Ukraine /ID# 209556, Kharkiv, Kharkivs’ka Oblast’
  - Scientific Research Institute of Invalid Rehabilitation /ID# 207873, Vinnytsia, Vinnytsia Oblast
  - CNE Cherkasy Regional Hospital of Cherkasy Regional Council /ID# 207912, Cherkasy
  - MNPE Chernihiv Regional Hospital of the Chernihiv Region Council /ID# 207730, Chernihiv
  - PNE City Multifunctional Hospital No.18 /ID# 207911, Kharkiv
  - Khmelnytskyi Regional Hospital /ID# 207753, Khmelnytskyi
  - MI Kryvyi Rih City Clinical Hospital No.2 /ID# 207748, Kryvyi Rih
  - Medical Center OK Clinic /ID# 207749, Kyiv
  - Communal Enterprise Volyn Regional Clinical hospital of the Volyn Regional Coun /ID# 208276, Lutsk
  - Lviv Municipal City Clinical Hospital #4 /ID# 207715, Lviv
  - PI "Poltava Regional Clinical Hospital n.a. M.V.Sklifosovsky" /ID# 207872, Poltava
  - Public Institution 6th City Clinical Hospital /ID# 207754, Zaporizhzhia
- United Kingdom (7):
  - Duplicate_Barts Health NHS Trust /ID# 210534, London, London, City of
  - NHS Greater Glasgow and Clyde /ID# 214942, Glasgow, Scotland
  - Midlands Partnership NHS Foundation Trust /ID# 214941, Stafford, Staffordshire
  - Manchester University NHS Foundation Trust /ID# 207928, Manchester
  - Duplicate_Wirral University Teaching Hospital NHS Foundation Trust /ID# 210535, Metropolitan Borough of Wirral
  - Portsmouth Hospitals University NHS Trust /ID# 207932, Portsmouth
  - Torbay and South Devon Nhs Foundation Trust /Id# 207931, Torquay

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Result] Kristensen LE, Keiserman M, Papp K, McCasland L, White D, Lu W, Wang Z, Soliman AM, Eldred A, Barcomb L, Behrens F. Efficacy and safety of risankizumab for active psoriatic arthritis: 24-week results from the randomised, double-blind, phase 3 KEEPsAKE 1 trial. Ann Rheum Dis. 2022 Feb;81(2):225-231. doi: 10.1136/annrheumdis-2021-221019. Epub 2021 Dec 15. PMID 34911706
- [Derived] Gossec L, Balanescu A, D'Agostino MA, Ogdie A, Sewerin P, Deng Y, Shi L, Sugimoto Y, Zhong S, Xing Y, Lippe R, Kishimoto M. Efficacy of Risankizumab across distinct PsA phenotypes identified with machine learning analytics using data from biologic DMARD-Naive patients in two phase 3 clinical trials. Arthritis Res Ther. 2025 Nov 29;28(1):2. doi: 10.1186/s13075-025-03670-0. PMID 41318485
- [Derived] Ostor A, Van den Bosch F, Papp K, Keiserman M, Blanco R, Crowley A, White D, Biljan A, Madihlaba T, Carter K, Liu F, Soliman AM, Ashley D, Chen M, Glotfelty L, Kivitz A. Efficacy and Safety of Risankizumab for Active Psoriatic Arthritis: 196-Week Results from the KEEPsAKE 1 and KEEPsAKE 2 Randomized Clinical Trials. Rheumatol Ther. 2025 Dec;12(6):1103-1123. doi: 10.1007/s40744-025-00793-3. Epub 2025 Sep 30. PMID 41028616
- [Derived] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Risankizumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Oct;11(5):1403-1412. doi: 10.1007/s40744-024-00706-w. Epub 2024 Aug 9. PMID 39120849
- [Derived] Kwatra SG, Khattri S, Amin AZ, Ranza R, Kaplan B, Shi L, Padilla B, Soliman AM, McGonagle D. Enthesitis and Dactylitis Resolution with Risankizumab for Active Psoriatic Arthritis: Integrated Analysis of the Randomized KEEPsAKE 1 and 2 Trials. Dermatol Ther (Heidelb). 2024 Jun;14(6):1517-1530. doi: 10.1007/s13555-024-01174-4. Epub 2024 May 13. PMID 38739215
- [Derived] Kristensen LE, Keiserman M, Papp K, McCasland L, White D, Carter K, Lippe R, Photowala H, Drogaris L, Soliman AM, Chen M, Padilla B, Behrens F. Efficacy and Safety of Risankizumab for Active Psoriatic Arthritis: 100-Week Results from the Phase 3 KEEPsAKE 1 Randomized Clinical Trial. Rheumatol Ther. 2024 Jun;11(3):617-632. doi: 10.1007/s40744-024-00654-5. Epub 2024 Mar 18. PMID 38498141
- [Derived] Kristensen LE, Keiserman M, Papp K, McCasland L, White D, Lu W, Soliman AM, Eldred A, Barcomb L, Behrens F. Efficacy and safety of risankizumab for active psoriatic arthritis: 52-week results from the KEEPsAKE 1 study. Rheumatology (Oxford). 2023 Jun 1;62(6):2113-2121. doi: 10.1093/rheumatology/keac607. PMID 36282530
- [Derived] Thakre N, D'Cunha R, Goebel A, Liu W, Pang Y, Suleiman AA. Population Pharmacokinetics and Exposure-Response Analyses for Risankizumab in Patients with Active Psoriatic Arthritis. Rheumatol Ther. 2022 Dec;9(6):1587-1603. doi: 10.1007/s40744-022-00495-0. Epub 2022 Sep 30. PMID 36178584
- [Derived] Kristensen LE, Soliman AM, Papp K, White D, Barcomb L, Lu W, Eldred A, Behrens F. Risankizumab improved health-related quality of life, fatigue, pain and work productivity in psoriatic arthritis: results of KEEPsAKE 1. Rheumatology (Oxford). 2023 Feb 1;62(2):629-637. doi: 10.1093/rheumatology/keac342. PMID 35801915
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M16-011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 186 sites in 38 countries globally. The study includes a 24-week double-blind placebo-controlled treatment period (Period 1) and an ongoing 184-week open-label treatment period (Period 2). Results are reported for Period 1 which was from 25 March 2019 to 8 October 2020.
Pre-assignment Details: Participants were randomized equally (1:1 ratio) to receive double-blind treatment with risankizumab 150 mg or matched placebo for 24 weeks. Randomization was stratified by extent of psoriasis (≥ 3% body surface area [BSA] or < 3% BSA), current conventional synthetic disease-modifying anti-rheumatic drug (csDMARD) use (0 vs ≥ 1), presence of dactylitis (yes vs no), and presence of enthesitis (yes vs no) at Baseline.
Groups:
- Placebo: Participants randomized to receive placebo administered by subcutaneous injection at Week 0, Week 4, and Week 16 in Period 1.
- Risankizumab: Participants randomized to receive 150 mg risankizumab administered by subcutaneous injection at Week 0, Week 4, and Week 16 in Period 1.
Period: Overall Study
Arm/Group | Placebo | Risankizumab
Started | 481 | 483
Completed (Completed Period 1 study participation) | 467 | 473
Not Completed | 14 | 10
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Lost to Follow-up | 3 | 0
Not completed — Lack of Efficacy | 1 | 1
Not completed — Coronavirus Disease-2019 (COVID-19) Logistical Restrictions | 1 | 2
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo: Participants received placebo administered by subcutaneous injection at Week 0, Week 4, and Week 16 in Period 1.
- Risankizumab: Participants received 150 mg risankizumab administered by subcutaneous injection at Week 0, Week 4, and Week 16 in Period 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | Risankizumab | Total
Number analyzed (Participants) | 481 | 483 | 964
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (12.10) | 51.3 (12.21) | 51.3 (12.15)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 408 | 414 | 822
  ≥ 65 years | 73 | 69 | 142
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 231 | 478
  Male | 234 | 252 | 486
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 92 | 93 | 185
  Not Hispanic or Latino | 389 | 390 | 779
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 451 | 454 | 905
  Black or African American | 2 | 4 | 6
  Asian | 22 | 13 | 35
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  American Indian or Alaska Native | 0 | 1 | 1
  Multiple | 5 | 8 | 13
Current Use of csDMARD [Count of Participants; unit: Participants]
  Yes | 364 | 366 | 730
  No | 117 | 117 | 234
Extent of Psoriasis [Count of Participants; unit: Participants] — The extent of psoriasis was measured by the physician as the total body surface area (BSA) involved with psoriasis. For purposes of clinical estimation, the total surface of the participant's palm and five digits was assumed to be approximately equivalent to 1% of BSA.
  Participants
    < 3% BSA | 209 | 210 | 419
    ≥ 3% BSA | 272 | 273 | 545
Presence of Dactylitis [Count of Participants; unit: Participants] — Dactylitis is characterized by swelling of the fingers or toes. The Leeds dactylitis index (LDI) basic is a score based on finger circumference and tenderness, assessed across all digits. The LDI basic measures the ratio of the circumference of the affected digit to the circumference of the digit on the opposite hand or foot, using a minimum difference of 10% to define a dactylitic digit. The ratio of circumference is multiplied by a tenderness score (1 for tender, 0 for non-tender). Scores for each digit are summed for the total LDI. The presence of dactylitis is defined as LDI > 0.
  Participants
    Yes | 147 | 148 | 295
    No | 334 | 335 | 669
Presence of Enthesitis [Count of Participants; unit: Participants] — Enthesitis is inflammation of the entheses, the specific point where tendons or ligaments attach to bone. The Leeds enthesitis index (LEI) is a validated enthesitis index that uses 6 sites for evaluation of enthesitis: lateral epicondyle humerus left and right, Achilles tendon insertion left and right and medial condyle femur left and right. Tenderness on examination is recorded as either present (1) or absent (0) for each of the 6 sites, for an overall score range of 0 - 6. Presence of enthesitis is defined as an LEI > 0.
  Participants
    Yes | 290 | 297 | 587
    No | 191 | 186 | 377
Tender Joint Count [Mean (Standard Deviation); unit: joints] — A total of 68 joints were assessed for the presence or absence of tenderness by pressure manipulation on physical examination.
  joints | 20.5 (12.79) | 20.8 (14.05) | 20.6 (13.43)
Swollen Joint Count [Mean (Standard Deviation); unit: joints] — A total of 66 joints were assessed for the presence or absence of swelling by directed physical examination.
  joints | 12.2 (8.02) | 12.1 (7.80) | 12.2 (7.91)
Patient's Assessment of Pain [Mean (Standard Deviation); unit: mm] — Participants were asked to indicate the severity of their arthritis pain within the previous 24 hours using a horizontal 100 mm visual analog scale (VAS), ranging from 0 (no pain) to 100 (severe pain). Population: Participants with available data
  mm
    number analyzed (Participants) | 479 | 482 | 961
    (all) | 57.1 (22.61) | 57.1 (22.57) | 57.1 (22.58)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — Participants were asked to rate their current psoriatic arthritis disease activity within the past 24 hours on a horizontal 100 mm VAS ranging from 0 (very well) to 100 (very poorly). Population: Participants with availabe data
  mm
    number analyzed (Participants) | 479 | 482 | 961
    (all) | 57.4 (22.06) | 57.9 (21.75) | 57.6 (21.89)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — The physician rated the participant's current global psoriatic arthritis disease activity in the past 24 hours (independently from the participant's assessment) on a 100 mm horizontal VAS ranging from 0 (very well) to 100 (very poorly). Population: Participants with available data
  mm
    number analyzed (Participants) | 461 | 466 | 927
    (all) | 62.4 (16.99) | 61.3 (17.64) | 61.8 (17.32)
Health Assessment Questionnaire Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: score on a scale] — The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. Population: Participants with available data
  score on a scale
    number analyzed (Participants) | 479 | 482 | 961
    (all) | 1.17 (0.651) | 1.15 (0.664) | 1.16 (0.658)
High-sensitivity C-reactive Protein (hsCRP) Level [Mean (Standard Deviation); unit: mg/L] | 11.33 (14.122) | 11.88 (15.933) | 11.60 (15.051)
Psoriasis Area Severity Index (PASI) Score [Mean (Standard Deviation); unit: score on a scale] — PASI is a composite score based on the percentage of the body surface area (BSA) affected by psoriasis and the intensity of erythema (reddening), induration, and desquamation of lesions assessed at 4 anatomic sites (head, upper extremities, trunk, and lower extremities). At each location, the percentage of BSA involvement is assigned a score from 0 (no involvement) to 6 (90% to 100% involvement), and erythema, induration, and desquamation are scored on a scale from 0 (no symptoms) to 4 (very marked). The PASI score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). Population: Participants with psoriasis BSA involvement ≥ 3% at Baseline
  score on a scale
    number analyzed (Participants) | 271 | 273 | 544
    (all) | 10.04 (10.436) | 10.89 (10.052) | 10.47 (10.244)
Modified Nail Psoriasis Severity Index (mNAPSI) Score [Mean (Standard Deviation); unit: score on a scale] — Fingernails were assessed for onycholysis (separation of the nail plate from the nail bed) and oil-drop dyschromia (reddish-brown discoloration under nail plate) on a scale of 0 (none) to 3 (>30% of nail), pitting on a scale of 0 (0 pits) to 3 (>50 pits), and nail plate crumbling on a scale of 0 (none) to 3 (>50% of nail crumbling) and absence/presence (0/1) of leukonychia (white spots), splinter hemorrhages, hyperkeratosis and red spots in the lunula. The mNAPSI score is the sum of all components for all fingernails and ranges from 0 (no nail psoriasis) to 130 (most severe nail psoriasis). Population: Participants with psoriatic nail disease at Baseline
  score on a scale
    number analyzed (Participants) | 338 | 309 | 647
    (all) | 16.56 (16.045) | 18.13 (16.443) | 17.31 (16.243)
Physician Global Assessment of Fingernail Psoriasis Score (PGA-F) [Mean (Standard Deviation); unit: score on a scale] — The PGA-F is a clinician-rated outcomes assessment used to measure the severity of signs and symptoms associated with fingernail psoriasis. Participant's fingernails were assessed separately for nail bed signs and nail matrix signs of disease on a scale from 0 (clear) to 4 (severe). A participant's overall global score is the worse of the nail bed score and nail matrix score. For example, if a participant had a nail bed score '2' and a nail matrix score of '4,' this participant's overall score was '4.' Population: Participants with psoriatic nail disease at Baseline
  score on a scale
    number analyzed (Participants) | 338 | 309 | 647
    (all) | 2.0 (1.00) | 2.1 (1.04) | 2.0 (1.02)
Short-Form 36 (SF-36) Physical Component Summary (PCS) Score [Mean (Standard Deviation); unit: score on a scale] — The SF-36 Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component summary is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The PCS ranges from 0 to 100, with a normative mean value of 50; higher scores are associated with less disability. Population: Participants with available data
  score on a scale
    number analyzed (Participants) | 477 | 482 | 959
    (all) | 35.15 (7.692) | 35.24 (8.094) | 35.20 (7.893)
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score [Mean (Standard Deviation); unit: score on a scale] — The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days, including physical fatigue, functional fatigue, emotional fatigue, and social consequences of fatigue. Participants respond to the questions on a scale from 0 (not at all) to 4 (very much). The FACIT-Fatigue score is computed by summing the item scores, after reversing items worded in the negative direction. The FACIT-Fatigue score ranges from 0 to 52, where higher scores represent less fatigue. Population: Participants with available data
  score on a scale
    number analyzed (Participants) | 477 | 482 | 959
    (all) | 29.3 (11.23) | 29.4 (11.28) | 29.4 (11.25)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 24
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 24
Population: Full analysis set; Non-responder imputation incorporating multiple imputation (MI) to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 481 | 483
percentage of participants | 33.5 [29.3 to 37.8] | 57.3 [52.9 to 61.8]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; The comparison between the risankizumab and placebo treatment groups for the primary efficacy endpoint (ACR20 at Week 24) was performed using the Cochran-Mantel-Haenszel (CMH) test adjusting for the stratification factors of baseline psoriasis (≥ 3%/< 3% body surface area), presence of dactylitis (yes/no), presence of enthesitis (yes/no) and current csDMARD use (0/≥ 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — All primary and ranked secondary efficacy endpoints were tested with multiplicity adjustment via a fixed sequence testing procedure to control the family-wise type I error rate at α=0.05 (two- sided); CMH test adjusted for the stratification factors of current csDMARD use, presence of dactylitis, enthesitis and extent of psoriasis at Baseline; Response Rate Difference = 24.0, 95% CI 2-sided [18.0 to 30.0] — Response Rate Difference = Risankizumab - Placebo

2. Secondary Outcome: Change From Baseline In Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 24
Description: The Health Assessment Questionnaire Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
  A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline and Week 24
Population: Full analysis set; a mixed effect model repeat measurement (MMRM) analysis with longitudinal data from observed cases up to Week 24, excluding data after initiation of rescue medication or initiation of concomitant medications for psoriatic arthritis (PsA) use that could meaningfully impact efficacy assessment, was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 479 | 482
score on a scale | -0.11 [-0.16 to -0.06] | -0.31 [-0.36 to -0.27]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; MMRM analysis including treatment, visit, treatment-by-visit interaction, and stratification factors as fixed factors and Baseline value as covariate; Least Squares (LS) Mean Difference = -0.20, 95% CI 2-sided [-0.26 to -0.14] — Difference = Risankizumab - Placebo

3. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 90 Response at Week 24
Description: PASI is a composite score based on the percentage of the body surface area (BSA) affected by psoriasis and the intensity of erythema (reddening), induration (thickening or hardening of the skin), and desquamation (peeling of the skin) of lesions assessed at 4 anatomic sites (head, upper extremities, trunk, and lower extremities). At each location, the percentage of BSA involvement is assigned a score from 0 (no involvement) to 6 (90% to 100% involvement), and erythema, induration, and desquamation are scored on a scale from 0 (no symptoms) to 4 (very marked).
  The PASI score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). A PASI 90 response is the percentage of participants who achieved at least a 90% reduction (improvement) from Baseline in PASI score.
Time Frame: Baseline and Week 24
Population: Full analysis set participants with Baseline psoriasis BSA involvement ≥ 3%; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 272 | 273
percentage of participants | 9.9 [6.4 to 13.5] | 52.3 [46.4 to 58.3]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 42.5, 95% CI 2-sided [35.6 to 49.3] — Response Rate Difference = Risankizumab - Placebo

4. Secondary Outcome: Percentage of Participants With an ACR20 Response at Week 16
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: Full analysis set; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 481 | 483
percentage of participants | 33.4 [28.9 to 37.9] | 56.3 [51.7 to 60.8]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 23.1, 95% CI 2-sided [16.8 to 29.4] — Response Rate Difference = Risankizumab - Placebo

5. Secondary Outcome: Percentage of Participants Achieving Minimal Disease Activity (MDA) at Week 24
Description: A participant was classified as achieving MDA if 5 of the following 7 criteria were met:
  * Tender joint count (out of 68 joints) ≤ 1
  * Swollen joint count (out of 66 joints) ≤ 1
  * PASI score ≤ 1 (score ranges from 0 - 72) or percent BSA involved with psoriasis ≤ 3%
  * Patient's assessment of pain ≤ 15 (VAS from 0 to 100)
  * Patient's Global Assessment of disease activity ≤ 20 (VAS from 0 to 100)
  * HAQ-DI score ≤ 0.5 (index score ranges from 0 to 3)
  * Leeds Enthesitis Index ≤ 1 (assesses the presence or absence of enthesitis at 3 bilateral sites, for an overall score range from 0 to 6)
Time Frame: Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 481 | 483
percentage of participants | 10.2 [7.5 to 12.9] | 25.0 [21.2 to 28.9]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 14.8, 95% CI 2-sided [10.2 to 19.4] — Response Rate Difference = Risankizumab - Placebo

6. Secondary Outcome: Change From Baseline in Modified Nail Psoriasis Severity Index (mNAPSI) Score at Week 24
Description: The investigator assessed each fingernail for onycholysis (separation of the nail plate from the nail bed) and oil-drop (salmon patch) dyschromia (reddish-brown discoloration under the nail plate) on a scale of 0 (none present) to 3 (>30% of the nail), pitting (small, sharply defined depressions in the nail surface) on a scale of 0 (0 pits present) to 3 (> 50 pits present), and nail plate crumbling on a scale of 0 (no crumbling) to 3 (>50% of nail has crumbling) and presence (1) or absence (0) of leukonychia (white spots), splinter hemorrhages, nail bed hyperkeratosis, and red spots in the lunula.
  The mNAPSI score is calculated as the sum of all the components for all of the participant's fingernails giving a range of possible scores from 0 (absence of nail psoriasis) to 130 (the most severe nail psoriasis). A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: Full analysis set with nail psoriasis at Baseline; a mixed effect model repeat measurement analysis with longitudinal data from observed cases up to Week 24, excluding data after initiation of rescue medication or initiation of concomitant medications for psoriatic arthritis use that could meaningfully impact efficacy assessment, was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 338 | 309
score on a scale | -5.57 [-6.70 to -4.44] | -9.76 [-10.95 to -8.58]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -4.19, 95% CI 2-sided [-5.70 to -2.68] — Difference = Risankizumab - Placebo

7. Secondary Outcome: Change From Baseline in Fingernail-Physician Global Assessment (PGA-F)
Description: The PGA-F is a clinician-rated outcomes assessment used to measure the severity of signs and symptoms associated with fingernail psoriasis. Participant's fingernails were assessed separately for nail bed signs and nail matrix signs of disease on a scale from 0 (clear) to 4 (severe). A participant's overall global score is the worse of the nail bed score and nail matrix score. For example, if a participant had a nail bed score '2' and a nail matrix score of '4,' this participant's overall score was '4.' A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 338 | 309
score on a scale | -0.4 [-0.5 to -0.3] | -0.8 [-1.0 to -0.7]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.6 to -0.3] — Difference = Risankizumab - Placebo

8. Secondary Outcome: Percentage of Participants With Resolution of Enthesitis at Week 24
Description: Resolution of enthesitis is defined as a Leeds Enthesitis Index (LEI) score = 0.
  LEI is an enthesitis measure developed specifically for PsA and assesses the presence or absence of tenderness at the following 3 bilateral enthesial sites: medial femoral condyles, lateral epicondyles of the humerus, and Achilles tendon insertions. Tenderness on examination is recorded as either present (coded as 1), absent (coded as 0), or not assessed for each of the 6 sites. The LEI is calculated by taking the sum of the scores from the 6 sites. The LEI ranges from 0 to 6 (worst).
  To increase the sample size due to the smaller number of participants with enthesitis at Baseline, the pre-specified analysis of the resolution of enthesitis included pooled data from KEEPsAKE 1 (this study) and the companion study KEEPsAKE 2 (M15-998; NCT03671148).
Time Frame: Week 24
Population: Full analysis set participants with a Baseline LEI > 0; Includes pooled data from KEEPsAKE 1 (this study) and the companion study M15-998 (NCT03671148; KEEPsAKE2). Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 448 | 444
percentage of participants | 34.8 [30.4 to 39.2] | 48.4 [43.8 to 53.1]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; The pre-specified analysis for the resolution of enthesitis included pooled data from KEEPsAKE 1 (this study) and KEEPsAKE 2 (M15-998; NCT03671148); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; CMH test adjusted for the stratification factors of current csDMARD use and extent of psoriasis at Baseline and study; Response Rate Difference = 13.9, 95% CI 2-sided [7.6 to 20.2] — Response Rate Difference = Risankizumab - Placebo

9. Secondary Outcome: Percentage of Participants With Resolution of Dactylitis at Week 24
Description: Resolution of dactylitis is defined as a Leeds Dactylitis Index (LDI) score = 0.
  LDI basic is a score based on finger circumference and tenderness, assessed across all digits. The LDI basic measures the ratio of the circumference of the affected digit to the circumference of the digit on the opposite hand or foot, using a minimum difference of 10% to define a dactylitic digit. The ratio of circumference is multiplied by a tenderness score (1 for tender, 0 for non-tender). If both sides of a digit are considered involved, or the circumference of the contralateral digit cannot be obtained, a standard reference table is used. Scores from each digit are summed to provide the final LDI. A higher LDI indicates worse dactylitis.
  To increase sample size due to the smaller number of participants with dactylitis at Baseline, the pre-specified analysis of the resolution of dactylitis included pooled data from KEEPsAKE 1 (this study) and the companion study KEEPsAKE 2 (M15-998; NCT03671148).
Time Frame: Week 24
Population: Full analysis set participants with a Baseline LDI > 0; Includes pooled data from KEEPsAKE 1 (this study) and the companion study M15-998 (NCT03671148; KEEPsAKE2). Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 204 | 188
percentage of participants | 51.0 [44.1 to 57.8] | 68.1 [61.4 to 74.7]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; The pre-specified analysis for the resolution of dactylitis included pooled data from KEEPsAKE 1 (this study) and KEEPsAKE 2 (M15-998; NCT03671148); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; CMH test adjusted for the stratification factors of current csDMARD use, extent of psoriasis at Baseline, and study; Response Rate Difference = 16.9, 95% CI 2-sided [7.5 to 26.4] — Response Rate Difference = Risankizumab - Placebo

10. Secondary Outcome: Change From Baseline in PsA Modified Total Sharp Score (mTSS) at Week 24
Description: The Sharp-van der Heijde modified scoring method for PsA measures the level of joint damage from radiographs of the hands and feet, and was assessed by 2 independent, blinded readers.
  Joint erosion severity was assessed in 20 joints in each hand and wrist and 6 joints in each foot. Each joint was scored from 0 (no erosion) to 5 for hands/wrists or to 10 for feet (complete collapse). The total erosion score ranges from 0 to 320 (worst).
  Joint space narrowing (JSN) was assessed in 20 joints of each hand and wrist, and 6 joints of each foot, from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation). The total JSN score ranges from 0 to 208 (worst).
  Joints with gross osteolysis or pencil in cup were assigned the maximum score for both erosions and JSN.
  The total mTSS score is the sum of the joint erosion and JSN scores and ranges from 0 (normal) to 528 (worst).
Time Frame: Baseline and Week 24
Population: Full analysis set participants with available data at Baseline; linear extrapolation was used for participants who discontinued prior to Week 24 or who were rescued prior to Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 457 | 458
score on a scale | 0.32 [0.11 to 0.53] | 0.23 [0.02 to 0.44]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p = 0.496, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model including treatment and the stratification factors and baseline value as covariates; LS Mean Difference = -0.09, 95% CI 2-sided [-0.36 to 0.17] — Difference = Risankizumab - Placebo

11. Secondary Outcome: Change From Baseline In 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score at Week 24
Description: The Short Form 36-Item Health Survey (SF-36) Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component summary is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The SF-36 PCS ranges from 0 to 100. A linear algorithm was applied to the calculation of the PCS which has a normative mean value of 50. Higher scores are associated with less disability; a score of 100 is equivalent to no disability and a score of 0 is equivalent to maximum disability. A positive change from Baseline score indicates improvement.
Time Frame: Baseline and Week 24
Population: Full analysis set; a mixed effect model repeat measurement analysis with longitudinal data from observed cases up to Week 24, excluding data after initiation of rescue medication or initiation of concomitant medications for psoriatic arthritis use that could meaningfully impact efficacy assessment, was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 477 | 482
score on a scale | 3.20 [2.50 to 3.89] | 6.52 [5.83 to 7.20]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Other; p < 0.001, Mixed Effect Model Repeated Measurement — This comparison was not tested for statistical significance because the hierarchical testing procedures stopped at the change from Baseline in PsA-mTSS comparison; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 3.32, 95% CI 2-sided [2.42 to 4.22] — Difference = Risankizumab - Placebo

12. Secondary Outcome: Change From Baseline In Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 24
Description: The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days, including physical fatigue (e.g., I feel tired), functional fatigue (e.g., trouble finishing things), emotional fatigue (e.g., frustration), and social consequences of fatigue (e.g., limits social activity). Participants respond to the questions on a scale from 0 (not at all) to 4 (very much).
  The FACIT-Fatigue score is computed by summing the item scores, after reversing those items that are worded in the negative direction. The FACIT-Fatigue score ranges from 0 to 52, where higher scores represent less fatigue.
  A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: Full analysis set; a mixed effect model repeat measurement analysis with longitudinal data from observed cases up to Week 24, excluding data after initiation of rescue medication or initiation of concomitant medications for psoriatic arthritis (PsA) use that could meaningfully impact efficacy assessment, was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 477 | 482
score on a scale | 3.9 [3.1 to 4.7] | 6.5 [5.6 to 7.3]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Other; p < 0.001, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 2.6, 95% CI 2-sided [1.5 to 3.7] — Difference = Risankizumab - Placebo

13. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 24
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 481 | 483
percentage of participants | 11.3 [8.4 to 14.1] | 33.4 [29.2 to 37.7]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 22.2, 95% CI 2-sided [17.3 to 27.2] — Response Rate Difference = Risankizumab - Placebo

14. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 24
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 481 | 483
percentage of participants | 4.7 [2.8 to 6.7] | 15.3 [12.0 to 18.5]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 10.5, 95% CI 2-sided [6.9 to 14.2] — Response Rate Difference = Risankizumab - Placebo

ADVERSE EVENTS:
Time Frame: From first dose of study drug to Week 24
Arm/Group | Placebo | Risankizumab
All-Cause Mortality (participants affected / at risk) | 0/481 | 1/483
Serious Adverse Events (participants affected / at risk) | 18/481 | 12/483
Other Adverse Events (participants affected / at risk) | 0/481 | 0/483
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=481) | Risankizumab (N=483)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
BLOOD LOSS ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
APPENDICITIS PERFORATED (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (2) | 1 (1)
COMPLICATED APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
DYSENTERY (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
ORAL BACTERIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
URETEROCELE (Renal and urinary disorders) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (3):
  • Study Protocol (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT03675308/Prot_001.pdf
  • Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT03675308/SAP_002.pdf
  • Informed Consent Form (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT03675308/ICF_000.pdf